CLINICAL TRIAL: NCT06105190
Title: Prospective, Multicenter, Controlled, Randomized, Masked Study to Evaluate the Safety and Performance of LuxSmart IOL as Compared With LuxGood IOL In Subjects Undergoing Cataract Extraction
Brief Title: Clinical Study to Evaluate Clinical Outcomes of LuxSmart IOL as Compared With LuxGood IOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cutting Edge SAS (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE2201
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular Lens; IOL; hydrophobic; EDOF
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is planned as a double-masked study. The subjects will not be informed about the implanted lens before exiting the study. Only the investigator implanting the lens as well as one administrative person will know about the arm, the subject is assigned to. Outcome assessors will not be able to receive information about the implanted lens. Data analyst will get to know about the patient assignment after data evaluation only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): Experimental arm: Premium monofocal intraocular lens LuxSmart
  Interventions: Device: Implantation of premium monofocal IOL, LuxSmart (device under investigation)
- IOL implantation active comparator (Active Comparator): Comparator arm: Monofocal intraocular lens LuxGood
  Interventions: Device: Implantation of monofocal IOL, LuxGood (control device)

INTERVENTIONS:
Device: Implantation of premium monofocal IOL, LuxSmart (device under investigation) — Patients will be implanted with study IOL in both eyes
  Arms: IOL implantation experimental
Device: Implantation of monofocal IOL, LuxGood (control device) — Patients will be implanted with Control IOL in both eyes
  Arms: IOL implantation active comparator

SUMMARY:
This study is a multicentric, prospective, randomised, controlled, post-market clinical follow up (PMCF) study to investigate safety, visual outcomes and contrast sensitivity after bilateral implantation of either LuxSmart IOLs (study group) or LuxGood IOLs (control group).

DETAILED DESCRIPTION:
This study is a multicentric, prospective, randomised, controlled, post-market clinical follow up (PMCF) study whereby subjects undergoing routine cataract surgery will have bilateral implantation of either LuxSmart IOLs (study group) or LuxGood IOLs (control group).

The subjects will be randomized in a 1:1 ratio to receive the study or control lenses.

Both study and control IOLs, are CE approved The study and control IOLs, and all devices used for the study examinations, will be used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the subject.

The study device (LuxSmart) is a hydrophobic, premium monofocal intraocular lens (IOL) manufactured by the sponsor of this study. The control lens (LuxGood) is the monofocal parent lens sharing the same material and optic design but with slight differences in the optic design. The IOLs will be implanted as part of the routine cataract surgery on subjects suffering from cataract. The targeted study cohort represents the standard subject cohort for cataract surgery.

In total 238 subjects will be enrolled for this clinical study and receive bilateral implantation of the study or control lens based on a 1:1 randomization given by the EDC.

Subjects participating in the trial will attend a total of 6 to 10 study visits (1 preoperative, 1 or 2 operative and 4 - 7 postoperative visits that may be carried out at the same day if requirements allow) over a period of 6 months.

Data analyses will be performed after the last patient finished the 120-180 days postoperative examination.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically documented age-related cataracts in both eyes;
2. Calculated IOL power performed using an optical biometer is within the range of the study and control IOLs (15D to 28D);
3. Male or female adults aged 22 years or older on the day of first-eye surgery;
4. Regular corneal astigmatism ≤ 1.0 D (measured by IOL Master) in both eyes;
5. Clear intraocular media other than cataract in both eyes;
6. Willing and able to comply to the study requirements;
7. Capability to understand and sign an IRB approved informed consent form and privacy authorization;
8. Monocular best corrected visual acuity projected to be ≤ 0.18 logMAR (≥ 20/30 in Snellen) after IOL implantation in both eyes;
9. Subjects must have discontinued use of contact lenses for at least two weeks (for hard or toric lenses) or 3 days (for soft non-toric contact lenses) prior to the pre-operative examination, and throughout the clinical study;
10. Current contact lens wearers must demonstrate a stable refraction (within ±0.5 D for both sphere and cylinder) in each eye, as determined by distance manifest refraction on two consecutive examination dates after discontinuation of contact lens wear;

Exclusion Criteria:

1. Regular corneal astigmatism >1.0 D (measured by IOL Master) in one or both eyes;
2. Irregular astigmatism (measured by a topographer) in both eyes;
3. Difficulties for cooperation;
4. Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity loss to 20/30 or worse in one or both eyes;
5. Subjects with AMD suspicious eyes as determined by OCT examination;
6. Previous intraocular or corneal surgery in one or both eyes;
7. Traumatic cataract in one or both eyes as judged by investigator;
8. History or presence of macular edema in one or both eyes;
9. Instability of keratometry or biometry measurements; Acceptable maximum standard deviation: AL: ± 150 µm; ACD: ± 150 µm; K1 / K2: ± 0.15 D in both eyes;
10. Clinically significant, uncontrolled glaucoma with expected negative impact on Contrast Sensitivity and / or visual acuity outcomes in one or both eyes;
11. Pupil abnormalities (non-reactive, tonic, abnormally shaped) in one or both eyes;
12. Subjects that cannot achieve a minimum pharmacologic pupilar dilatation of 5 mm in one or both eyes;
13. Complicated surgery expected;
14. Ocular surface disease (clinical symptoms) in one or both eyes;
15. Clinically significant dry eye as determined by the investigator's judgement in one or both eyes;
16. Anterior segment pathology that might increase intraoperative risk or compromise IOL stability;
17. Diabetic retinopathy;
18. Congenital ocular anomalies;
19. Chronic or recurrent inflammatory eye diseases;
20. Active infectious conjunctivitis, keratitis or uveitis in either eye within 30 days prior to surgery;
21. Subjects who may be expected to require a combined or other surgical procedure in either eye;
22. Pregnant, lactating or, if able to bear children, unwilling to use medically acceptable birth control over the course of the study;
23. Concurrent or previous (within 30 days) participation in another drug or device investigation;
24. Systemic medications that may confound the outcome or increase the risk to the subject in the opinion of the investigator (tamsulosin hydrochloride (Flomax) or other medications with similar side effects (floppy iris syndrome);
25. Subjects with conditions that increase the risk of zonular rupture during cataract extraction procedure that may affect the postoperative centration or tilt of the lens;
26. Subjects who are expected to require retinal laser treatment;
27. Patients showing contraindications as listed in the current Instructions for use (IFU);
28. Unsuitable for study participation for any other reason, as determined by Investigator's clinical judgment (reason to be documented on eCRF).

In addition to above mentioned in- and exclusion criteria, subjects shall be discontinued when certain conditions are present at the time of surgery, including:

* zonular instability;
* need for iris manipulation;
* capsular fibrosis or other opacity; and
* inability to fixate IOL in desired position. In such cases, the subject shall be followed until the condition has stabilized.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Mean Corrected Distance Visual Acuity | 120-180 days postoperative
  The primary safety endpoint is to show that the mean monocular Corrected Distance Visual Acuity (CDVA) at at 120-180 days postoperative is statistically non-inferior to outcomes obtained in the control group using a non-inferiority margin of 0.1 logMAR, a 1-sided test and a significance level of 0.05. This analysis will be done for first implanted eyes as well as all implanted eyes per subject.
Co-Primary Safety Endpoint: Monocular Contrast Sensitivity - Between-group mean difference | 120-180 days postoperative
  The co-primary safety endpoint is to compare the outcomes on monocular contrast sensitivity under mesopic light conditions (with and without glare) between the study and the control group at 120-180 days postoperative. This analysis will be done for first implanted eyes per subject.
  The following Log Contrast Sensitivity Analysis will be performed:
  - Between-group mean difference in log contrast sensitivity with 90% non-parametric confidence interval for each spatial frequency.
Co-Primary Safety Endpoint: Monocular Contrast Sensitivity - descriptive statistics | 120-180 days postoperative
  The co-primary safety endpoint is to compare the outcomes on monocular contrast sensitivity under mesopic light conditions (with and without glare) between the study and the control group at 120-180 days postoperative. This analysis will be done for first implanted eyes per subject.
  The following Log Contrast Sensitivity Analysis will be performed:
  - Provide descriptive statistics for the log contrast sensitivity for each group (mean, SD, median, 0th, 25th, 50th 75th, and 100th percentiles) and for each spatial frequency.
Co-Primary Safety Endpoint: Monocular Contrast Sensitivity - frequency with glare | 120-180 days postoperative
  The co-primary safety endpoint is to compare the outcomes on monocular contrast sensitivity under mesopic light conditions with glare between the study and the control group at 120-180 days postoperative. This analysis will be done for first implanted eyes per subject.
  The following Log Contrast Sensitivity Analysis will be performed:
  - The percentage of eyes that can and cannot see the reference pattern for each spatial frequency.
Co-Primary Safety Endpoint: Monocular Contrast Sensitivity - frequency without glare | 120-180 days postoperative
  The co-primary safety endpoint is to compare the outcomes on monocular contrast sensitivity under mesopic light conditions without glare between the study and the control group at 120-180 days postoperative. This analysis will be done for first implanted eyes per subject.
  The following Log Contrast Sensitivity Analysis will be performed:
  - The percentage of eyes that can and cannot see the reference pattern for each spatial frequency.
Co-Primary Safety Endpoint: Best Corrected Distance Visual Acuity compared to historical data | 120-180 days postoperative
  The objective is to compare best corrected distance visual acuities (CDVA) above defined thresholds of the investigational product to the normative data stated in the according ISO norm (EN ISO 11979-7:2018) for posterior chamber intraocular lenses.
Co-Primary Safety Endpoint: Rates of Adverse Events | 120-180 days postoperative
  The objective is to compare the SPE (Safety and Performance Endpoints) rates of the investigational product to reference data stated in the according ISO standard for posterior intraocular lenses (EN ISO 11979-7:2018) based on minimum 100 subjects.
Co-Primary Safety Endpoint: Incidence of all SAE | 120-180 days postoperative
  The incidence of all Serious Adverse Events, including Secondary Surgical Interventions (SSIs) related to the optical properties of the IOL, in first-implanted eyes as well as all implanted eyes will be collected through Post-Operative Visit 4 (120 to 180 days after first and second eye implantation).
  The proportion of first implanted eyes and all implanted eyes with at least one serious adverse event will be summarized using categorical summary statistics by treatment received. Each eye will be counted only once in the calculation of the rate.
  There is no statistical hypothesis associated with the proportion of first implanted eyes with at least one serious adverse event.
Co-Primary Safety Endpoint: Rate of SSI Related to Optical Properties of the IOL | 120-180 days postoperative
  The rate of SSIs related to the optical properties of the IOL for first-implanted eyes as well as all implanted eyes will be reported through 120 to 180 days after first and second eye implantation.
  Secondary surgical interventions related to the optical properties of the IOL will be defined as IOL explantation, replacement, or repositioning due to subject intolerance of visual symptoms not adequately improved by spectacle correction. Each eye will be classified as either having undergone a secondary surgical intervention related to the optical properties of the IOL or not having undergone such an intervention. Secondary surgical interventions related to the optical properties of the IOL will be summarized categorically (Yes, No) by actual treatment received in a table.
Primary Performance Endpoint: Mean Distance Corrected Intermediate Visual Acuity | 120-180 days postoperative
  The primary efficacy endpoint is to show that the monocular Distance Corrected Intermediate Visual Acuity (DCIVA) at 120-180 days postoperative is statistically superior to outcomes obtained in the control group (1 sided test using significance of 0.025). To avoid bias, only the first implanted eye per subject will be considered for this calculation.
Co-Primary Performance Endpoint: Cumulative Distance Corrected Intermediate Visual Acuity | 120-180 days postoperative
  One co-primary efficacy endpoint is to show that the outcomes of the study device on monocular Distance Corrected Intermediate Visual Acuity (DCIVA) at 66 cm at 120-180 days postoperative needs to have at least 50% of eyes achieving 0.2 logMAR or better. To avoid bias, only the first implanted eye per subject will be considered for this calculation.
Co-Primary Performance Endpoint: Monocular best-corrected distance defocus | 120-180 days postoperative
  Monocular best-corrected distance defocus testing will be performed. The defocus range where the mean visual acuity of 0.2 logMAR or better is achieved will be derived by visual inspection of the mean defocus curve. The monocular depth of focus is defined as the defocus range from zero to the first negative vergence level, where the visual acuity is 0.2 logMAR or less.
  One co-primary efficacy endpoint is to show that the monocular depth of focus for the eyes implanted with the study device is at least 0.5 D greater than the depth of focus for the eyes implanted with the control device at 0.2 logMAR.

SECONDARY OUTCOMES:
Secondary Safety Endpoint: Best Corrected Distance Visual Acuity compared to historical data | 120-180 days postoperative
  The objective is to compare best corrected distance visual acuities (CDVA) above defined thresholds of the investigational product to the normative data stated in the according ISO norm (EN ISO 11979-7:2018) for posterior chamber intraocular lenses.
Secondary Performance Endpoint: Distance Corrected Near Visual Acuity (DCNVA) | 120-180 days postoperative
  Secondary performance endpoint is to show a statistically significant increase between pre-and postoperative findings on monocular Distance Corrected Near Visual Acuity (DCNVA) under photopic light conditions on the first implanted eye.
Secondary Performance Endpoint: Distance Corrected Intermediate Visual Acuity (DCIVA) | 120-180 days postoperative
  Secondary performance endpoint is to show a statistically significant increase between pre-and postoperative findings on monocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic light conditions on the first implanted eye.

OTHER OUTCOMES:
Binocular best-corrected distance defocus | 120-180 days postoperative
  In addition to the co-primary study endpoint on monocular defocus, binocular best-corrected distance defocus testing will be performed. The defocus range where the mean visual acuity of 0.2 logMAR or better is achieved will be derived by visual inspection of the mean defocus curve.
  The monocular depth of focus for the eyes implanted with the study device needs to be at least 0.5 D greater than the depth of focus for the eyes implanted with the control device at 0.2 logMAR [4].
  All measured outcomes data will be statistically compared to outcomes obtained in the control group.
Manifest refraction | Preoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The manifest refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2018. This data will also be used to calculate the manifest refractive spherical equivalent (MRSE)
Adjusted Mean Refractive Spherical Equivalent (MRSE) | 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The predictability of the postoperative manifest refraction will be evaluated using the absolute value of the adjusted MRSE calculated by the following formula:
  MRSEadjusted = MRSEpostop - MRSEtarget.
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | Preoperative, 1-2 days postoperative; 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular UDVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 4m distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 120-180 days postoperative
  Binocular UDVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 4m distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | Preoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular CDVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Monocular Corrected Distance Visual Acuity (low contrast CDVA) using low contrast (10%) optotypes under photopic light conditions | 120-180 days postoperative
  Monocular CDVA using low contrast (10%) optotypes is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions. This test is performed using a low-contrast acuity chart with 10% contrast (using the Weber definition: [background - optotype]/background).
Binocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 120-180 days postoperative
  Binocular CDVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Uncorrected Intermediate Visual Acuity (UIVA) under photopic light conditions | 30-60 days postoperative, 120-180 days postoperative
  Monocular UIVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 66cm distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity (UIVA) under photopic light conditions | 120-180 days postoperative
  Binocular UIVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 66cm distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Binocular Uncorrected Near Visual Acuity (UNVA) under photopic light conditions | 120-180 days postoperative
  Binocular UNVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 40cm distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic light conditions | 30-60 days postoperative, 120-180 days postoperative
  Monocular DCIVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) under mesopic light conditions | 120-180 days postoperative
  Monocular DCIVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under mesopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity (low contrast DCIVA) using low contrast (10%) optotypes under photopic light conditions | 120-180 days postoperative
  Monocular DCIVA using low contrast (10%) optotypes is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 66cmm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions. This test is performed using a low-contrast acuity chart with 10% contrast (using the Weber definition: [background - optotype]/background).
Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic light conditions | 120-180 days postoperative
  Binocular DCIVA is measured using the Clinical Trial Suite (M&S Technologies, Niles, USA) placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Binocular Distance Corrected Near Visual Acuity (DCNVA) under photopic light conditions | 120-180 days postoperative
  Binocular DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Subject Symptom Assessment | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Subject ocular and visual symptoms are collected at each postoperative visit through the use of non-directed questions. Responses will be recorded and characterized by severity (mild, moderate, severe) and divided into distinct groups of symptoms (halo, glare, ocular pain, ocular dryness, other).
  The percentage of eyes with ocular and visual symptoms will be reported divided into the mentioned severity levels and symptom groups. No scoring or scaling is used for this type of symptom assessment. All data obtained in the study group will be statistically compared to outcomes obtained in the control group.
Patient reported outcomes - Quality of Vision questionnaire | 30-60 days postoperative, 120-180 days postoperative
  To assess the subjective perception of disturbances by photic phenomena, the validated and verified Quality of Vision (QoV) questionnaire will be used.
  This questionnaire is a linear-scaled 30-item instrument and is designed with 10 symptoms rated in each of three scales (frequency, severity, and bothersome). Each of the three scales provides 4 answer options with the first answer being the best outcome and the 4th answer being the worst outcome:
  * Frequency answer options: never, occasionally, quite often, very often;
  * Severity answer options: not at all, mild, moderate, severe;
  * bothersome answer options: not at all, a little, quite, very.
  Based on the given answers, a QoV score in terms of symptom frequency, severity, and bothersome is calculated. The score ranges from 0 to 100 with 100 being the worst possible outcome.
Patient reported outcomes - Catquest-9SF 2011 questionnaire | 30-60 days postoperative, 120-180 days postoperative
  To assess if difficulties in daily life occur due to impaired sight. This questionnaire is a 9-item Rasch-scaled instrument to assess subjective perception of visual impairment after surgery.
  Each item has 4 answer options ranging from 'Yes, very great difficulty' to 'No, no difficulty'. with first answer being the best outcome and the last answer being the worst outcome. In addition, the subjects can state, that they cannot decide on the answer.
  The percentage of subjects per item will be reported per answer option. No scoring or scaling is used for this type of symptom assessment. All data obtained in the study group will be statistically compared to outcomes obtained in the control group.
Pupil Size under photopic light conditions | preoperative, 120-180 days postoperative
  Photopic pupil diameters are measured with a ruler allowing for a precision of at least +/-0.5 mm. In addition to the measurement with a ruler, pupil diameters under photopic light conditions will be recorded from the preoperative Pentacam measurement.
  For the photopic pupil diameters, eye illumination should be identical to that used for photopic contrast sensitivity testing. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 5 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Pupil Size under mesopic light conditions | preoperative, 120-180 days postoperative
  Mesopic pupil diameters are measured with a ruler allowing for a precision of at least +/-0.5 mm. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 5 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus examination with dilated pupil | preoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Corneal status | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Slitlamp examination - Iris status | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Iris Status
Slitlamp examination - Signs of inflammation | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  * Signs of inflammation
  * Anterior chamber cells,
  * Anterior chamber flare,
  * Cystoid macular oedema,
  * Hypopyon, and
  * Endophthalmitis.
Slitlamp examination - Pupillary block | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Pupillary block.
Slitlamp examination - Retinal detachment | preoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Retinal detachment.
Slitlamp examination - Status of anterior and posterior capsule | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Status of anterior and posterior capsule.
Slitlamp examination - IOL decentration | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL decentration.
Slitlamp examination - IOL tilt | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL tilt.
Slitlamp examination - IOL discoloration | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL discoloration.
Slitlamp examination - IOL opacity | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL opacity.
Intraocular pressure (IOP) measurement | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Keratometry | Preoperative
  Keratometric measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power | during surgery
  The power of the implanted IOL will be recorded.
Target refraction | during surgery
  The target refraction given by the IOL calculator is recorded. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Preoperative
  An OCT (optical coherence tomography) image will be taken at the preoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Biometry | Preoperative
  Biometry measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Corneal topography | Preoperative
  Pentacam device (Oculus, Germany) will be used to perform corneal topography. This examination is needed to exclude patients showing an irregular corneal astigmatism.
Corneal aberrometry | Preoperative
  Pentacam device (Oculus, Germany) will be used to perform corneal aberrometry measurement. The following values will be evaluated in this study: Spherical aberrations, high order aberrations.
Halo and glare scores | 30-60 days postoperative
  A Halo and Glare simulator software (Eyeland Design Network GmbH, Germany) will be used to assess the subjective perception of photic phenomena. The patients will be asked to adjust the halo and glare level in a simulated image to the amount they perceive of such photic phenomena. The scaling ranges from 0 to 100 with 0 indicating no halo or glare and 100 being the worst outcome.
  All data obtained in the study group will be statistically compared to outcomes obtained in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Dick, Prof., Principal Investigator — Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH
Locations (8):
- Univ.-Klinik fuer Augenheilkunde und Optometrie, Vienna, Austria
- Czechia (2):
  - Gemini Eye Clinic Vyškov, Vyškov
  - Gemini Eye Clinic Zlín, Zlín
- Germany (2):
  - Augenklinik Ahaus, Ahaus
  - Univ.-Klinikum Knappschaftskrankenhaus Bochum, Bochum
- Asian Eye Institute, Makati City, Manila, Philippines
- Tan Tock Seng Hospital, Singapore, Singapore
- Hospital Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205
- [Background] Lundstrom M, Pesudovs K. Catquest-9SF patient outcomes questionnaire: nine-item short-form Rasch-scaled revision of the Catquest questionnaire. J Cataract Refract Surg. 2009 Mar;35(3):504-13. doi: 10.1016/j.jcrs.2008.11.038. PMID 19251145